CLINICAL TRIAL: NCT00273325
Title: Observational Study of the Immunogenicity of Heptavalent Pneumococcal Conjugate Vaccine in Very-low-birth-weight Infants
Brief Title: Immunogenicity of PCV-7 Vaccine in VLBW Infants
Acronym: PCV-7
Status: Completed | Type: Observational
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: NICHD-NRN-0031; UL1RR024128 (NIH); UL1RR024160 (NIH); UL1RR024982 (NIH); UL1RR025008 (NIH); UL1RR025744 (NIH); UL1RR025777 (NIH); M01RR016587 (NIH); M01RR000030 (NIH); M01RR000032 (NIH); M01RR000039 (NIH); M01RR000044 (NIH); M01RR000633 (NIH); M01RR000070 (NIH); M01RR007122 (NIH); U01HD036790 (NIH); U10HD021385 (NIH); U10HD021397 (NIH); U10HD027851 (NIH); U10HD027880 (NIH); U10HD034216 (NIH); U10HD040492 (NIH); U10HD040498 (NIH); U10HD040521 (NIH); U10HD040689 (NIH)
Record Dates: First submitted 2005-09-09; First posted 2006-01-09 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Pneumococcal Infections; Streptococcus Pneumoniae; Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature
Keywords: NICHD Neonatal Research Network; Very Low Birth Weight (VLBW); Extremely Low Birth Weight (ELBW); Prematurity; Pneumococcal Vaccines; Vaccines, Conjugate; Immunogenicity; Vaccine Response; Heptavalent pneumococcal conjugate vaccine (PCV-7); pneumococcal polysaccharide, type 6B; Pneumococcal polysaccharide, type 14; Pneumococcal polysaccharide, type 19F,; Pneumococcal polysaccharide, 23F; Pneumococcal polysaccharide, 18C; Pneumococcal polysaccharide, 4; Pneumococcal polysaccharide, 9V
MeSH Terms: conditions — Pneumococcal Infections; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum was separated from blood samples. After all study assays were completed on all subjects, if a subject's parents asked that his/her serum not be stored, the serum was destroyed. For subjects whose parents permit it, leftover serum was re-labeled with a new, randomly-generated unique de-identifier, linked only to the subject's gestational age, birth weight, and chronologic age at the time of sampling. The link to any other subject identifiers will then be destroyed. The serum will be stored indefinitely at the University of Rochester for other, non-genetic-testing-related research.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Premature infants are at a high risk for pneumonia. The PCV-7 vaccine effectively prevents the invasive disease from Streptococcus pneumoniae in full-term infants, but was not thoroughly studied in premature infants. This study evaluated the effectiveness and safety of the vaccine given in routine practice to very low birth weight infants, looking at blood antibody levels 4-6 weeks after the final vaccine dose, and adverse events, survival, infections, and neurodevelopmental outcomes at 18-22 months corrected age.

DETAILED DESCRIPTION:
Streptococcus pneumoniae causes an estimated 10-25% of all pneumonias in the United States, and is responsible for an estimated 40,000 deaths per year. Invasive pneumococcal disease has a peak incidence of 235/100,000 among children aged 6-11 months. Pneumococcal meningitis carries a higher risk of death (15%) or neurodevelopmental impairment (12-28%) than Hib or Neisseria meningitides.

Premature infants are at a higher risk for invasive disease with Streptococcus pneumoniae. The heptavalent pneumococcal-CRM197 conjugate vaccine (PCV-7) effectively prevents invasive pneumococcal disease in full-term infants, but was been incompletely studied in premature infants. The American Academy of Pediatrics (AAP) recommends that "prematurely born infants, including infants of low birth weight, should be immunized at the usual chronological age in most cases", but cautions that "some studies suggest a reduced immune response in very low-birth-weight infants (<1500 g)."

This observational study assessed the effectiveness of the PCV-7 vaccine to generate a sufficient immune response in a safe manner when given to very low birth weight (VLBW) infants in routine pediatric practice. We hypothesized that among VLBW infants, the frequency of estimated minimum protective antibody titers to PCV-7 (>=0.15 μg/mL) would decrease with decreasing birth weight.

Infants 501-1500g birth weight and <32 0/7 weeks gestational age were enrolled from nine NICHD Neonatal Research Network centers from 2004 to 2006. Enrollment was stratified by weight group to yield approximately 20 infants per 100g increments from 501-1500g birth weight whose primary PCV-7 series was initiated before 3 months and completed by 8 months after birth. The infants' primary providers gave PCV-7 vaccination at 2, 4, and 6 months after birth. Infants had a single 2-ml blood sample drawn 4-6 weeks following the third dose of PCV-7. Antibodies for each of the seven vaccine serotypes included in PCV-7 were measured by enzyme-linked immunosorbent assay. Children were followed until 18-22 months corrected age to assess survival, infection, and neurodevelopmental outcomes.

ELIGIBILITY:
Inclusion criteria

* Gestational age <32 0/7 weeks
* Included in Neonatal Research Network Generic Database
* Family has a telephone at home
* Anticipated availability for blood draw 4-6 weeks following 3rd vaccine dose
* Consent obtained before first dose of PCV-7 is given

Exclusion criteria

* Known immunodeficiency
* HIV exposure
* Parental non-consent
* Primary care pediatrician not willing to participate
* Enrollment in a conflicting trial
* Infant has not received first dose of PCV-7 vaccine by 3 months of age

Max Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants <1,500g birth weight who receive the 3-dose primary series of PCV-7 immunization by 3 months and complete it by 8 months postnatal age
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2004-07; Primary Completion 2007-07 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Serotype 6B pneumococcal capsular polysaccharide antibody >=0.15 μg/ml | 4-6 weeks following the third dose of PCV-7

SECONDARY OUTCOMES:
Pneumococcal capsular polysaccharide antibody >=0.15 μg/ml for the other six vaccine serotypes | 4-6 weeks following the third dose of PCV-7
Pneumococcal capsular polysaccharide antibodies >=1.0 μg/ml for all seven vaccine serotypes | 4-6 weeks following the third dose of PCV-7
Geometric mean titers of pneumococcal capsular polysaccharide antibody to the seven vaccine serotypes | 4-6 weeks following the third dose of PCV-7
Pneumococcal capsular polysaccharide antibodies >=0.15 μg/ml and >=1.0 μg/ml, and geometric mean titers of antibody, to the seven vaccine serotypes in children completing the primary series, regardless of postnatal age | 4-6 weeks following the third dose of PCV-7
Opsonization of 6B pneumococcal capsular polysaccharide plus 1 low immunogenicity, high prevalence serotype (e.g., 23F) among infants in the lowest quartile of antibody response | 4-6 weeks following the third dose of PCV-7
Effect of possible mediating variables on the achievement of levels of serotype 6B pneumococcal capsular polysaccharide antibody >=0.15 μg/ml | 4-6 weeks following the third dose of PCV-7
Effect of pneumococcal conjugate immunization status (complete & timely v. complete v. incomplete) on outcome (survival, serious infection, neurodevelopmental outcome) at 18-22 months corrected age in infants <=1000g | 18-22 months corrected age
Levels of antibody >=0.15 μg/ml and >=1.0 μg/ml to Hib polyribosylribitol | 4-6 weeks following the third dose of PCV-7
Avidity of antibody to Hib-PRP among infants in the lowest quartile of antibody response,regardless of postnatal or gestational age | 4-6 weeks following the third dose of PCV-7

CONTACTS AND LOCATIONS:
Overall Officials: Ronald N. Goldberg, MD, Principal Investigator — Duke University; Barbara J. Stoll, MD, Principal Investigator — Emory University; Abhik Das, PhD, Principal Investigator — RTI International; Krisa P. Van Meurs, MD, Principal Investigator — Stanford University; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Shahnaz Duara, MD, Principal Investigator — University of Miami; Carl T. D'Angio, MD, Principal Investigator — University of Rochester; Pablo J. Sanchez, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; T. Michael O'Shea, MD MPH, Principal Investigator — Wake Forest University; Seetha Shankaran, MD, Principal Investigator — Wayne State University
Locations (10):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Wayne State University, Detroit, Michigan
  - University of Rochester, Rochester, New York
  - Wake Forest University, Charlotte, North Carolina
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

REFERENCES:
- [Result] D'Angio CT, Heyne RJ, O'Shea TM, Schelonka RL, Shankaran S, Duara S, Goldberg RN, Stoll BJ, Van Meurs KP, Vohr BR, Das A, Li L, Burton RL, Hastings B, Phelps DL, Sanchez PJ, Carlo WA, Stevenson DK, Higgins RD; NICHD Neonatal Research Network. Heptavalent pneumococcal conjugate vaccine immunogenicity in very-low-birth-weight, premature infants. Pediatr Infect Dis J. 2010 Jul;29(7):600-6. doi: 10.1097/INF.0b013e3181d264a6. PMID 20234331
- [Result] Wynn JL, Li L, Cotten CM, Phelps DL, Shankaran S, Goldberg RN, Carlo WA, Van Meurs K, Das A, Vohr BR, Higgins RD, Stoll BJ, D'Angio CT. Blood stream infection is associated with altered heptavalent pneumococcal conjugate vaccine immune responses in very low birth weight infants. J Perinatol. 2013 Aug;33(8):613-8. doi: 10.1038/jp.2013.5. Epub 2013 Jan 31. PMID 23370608
- [Result] Ang JY, Lua JL, Asmar BI, Shankaran S, Heyne RJ, Schelonka RL, Das A, Li L, Jackson DM, Higgins RD, D'Angio CT; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Nasopharyngeal carriage of Streptococcus pneumoniae in very low-birth-weight infants after administration of heptavalent pneumococcal conjugate vaccine. Arch Pediatr Adolesc Med. 2010 Dec;164(12):1173-5. doi: 10.1001/archpediatrics.2010.233. No abstract available. PMID 21135351
- [Result] D'Angio CT, Murray TE, Li L, Heyne RJ, O'Shea TM, Schelonka RL, Shankaran S, Duara S, Goldberg RN, Stoll BJ, Stevenson DK, Vohr BR, Phelps DL, Carlo WA, Pichichero ME, Das A, Higgins RD; NICHD Neonatal Research Network. Immunogenicity of Haemophilus influenzae type b protein conjugate vaccines in very low birth weight infants. Pediatr Infect Dis J. 2013 Dec;32(12):1400-2. doi: 10.1097/01.inf.0000437263.04493.7c. No abstract available. PMID 24569312
- See also: NICHD Neonatal Research Network — https://neonatal.rti.org/